CLINICAL TRIAL: NCT05868824
Title: Dynamic Blood Inflammatory Profile in Atopic Dermatitis Patients
Brief Title: Dynamic Blood Inflammatory Profile in Atopic Dermatitis Patients (ADAMUNE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-AOIP-05
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Cohort (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample for assessing cytokines will be performed at baseline and at follow-up visit 3 months after initiation of treatment. The blood sample will be performed as part of blood tests done for standard AD follow up.

SUMMARY:
This is a prospective, single-center, class 2 study to better characterize the immune response in immune response in the blood of atopic dermatitis. Investigators are following in the referral center of Nice, 100 patients with atopic dermatitis. Investigators plan to include 30 patients. Blood samples will be collected to assess cytokine levels after non-specific immune stimulation. immune stimulation. Whole blood will be collected and stimulated with immune ligands (anti-CD3 T-cell stimulating ligands associated with Thymic Stromal LymphoPoietin (TSLP) or TLR agonist R848 7/8 agonist stimulating NK (natural killer) lymphocytes and promoting T cell response) on lyophilized freeze-dried spheres (LyoSphere, Qiagen) within 8 hours of blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years.
* Patient with clinically diagnosed atopic dermatitis according to the criteria of Hanifin and Rajka.
* Moderate to severe defined by an Investigator's Global Assessment ³3 and eligible to systemic treatment.
* If the subject is a woman of childbearing potential, she has a negative urine pregnancy test.
* Subject is non-pregnant, non-lactating and is not planning for pregnancy during the study period.
* Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair his/her evaluation or which exposes the subject to an unacceptable risk by study participation.
* Subject is able to comprehend and willing to sign an Informed Consent and/or Assent Form.
* Affiliation to a social security scheme.
* Signed informed consent

Exclusion Criteria:

* Vulnerable person: pregnant or nursing woman, minor, adult under guardianship or deprived of liberty
* Patient with an infection
* Patient with other systemic inflammatory disease
* Patient with anti-inflammatory or immunosuppressive therapy
* Patient with a contraindication to JAK inhibitors
* Participants in other clinical therapeutic studies involving a drug that may interfere with the present evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Compare the dynamic blood cytokines profile by stimulating blood with immune ligands | At baseline
  Cytokines dosage, measured by ELISA, in blood sample before and after in vitro stimulation with immune ligands at baseline. Responders are defined by an Investigator's Global Assessment score £ 1, and by 2 or more points improvement.
Compare the dynamic blood cytokines profile by stimulating blood with immune ligands | After 3 months
  Cytokines dosage, measured by ELISA, in blood sample before and after in vitro stimulation with immune ligands after 3 months of treatment. Responders are defined by an Investigator's Global Assessment score £ 1, and by 2 or more points improvement.

SECONDARY OUTCOMES:
Compare cytokine dosage according to the different phenotypes of patients with atopic dermatitis. | 6 months
  Cytokines dosage, measured by ELISA, in blood sample before and after in vitro stimulation with immune ligands according to clinical phenotypes: moderate, severe, very severe defined by SCORAD, ethnic origin, the presence of specific clinical signs (head and neck dermatitis, "dirty neck", orbital darkening, perleche, Herthoge sign, nummular eczema, hand eczema, keratosis pilaris) or the presence of atopic comorbidities (asthma, conjunctivitis, allergic rhinitis, food allergy) in untreated patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No